CLINICAL TRIAL: NCT06200987
Title: Planned Penile Vibratory Stimulation in the Prevention of Sexual Dysfunction and Urinary Incontinence After Radical Prostatectomy: a Randomized Controlled Study
Brief Title: Penile Vibratory Stimulation in the Prevention of Sexual Dysfunction and Urinary Incontinence After Radical Prostatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Helene Reif Andersen, PhD fellow, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ProVibrate
Record Dates: First submitted 2023-12-29; First posted 2024-01-11 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy; Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): The group randomized to use the vibrator for 9 months
  Interventions: Device: Penile vibrator
- Controls (No Intervention): Usual standard treatment

INTERVENTIONS:
Device: Penile vibrator — In addition to standard treatment with PDE5-inhibitors the intervention is daily stimulation for five minutes with the vibrator for 9 months
  Arms: Intervention

SUMMARY:
To investigate if post-operative penile vibration stimulation kan be used to reduce or prevent sexual dysfunction and urinary incontinence after radical prostatectomy. This will be done in a randomized, controlled, non-blinded study. Men that undergo nerve preserving surgery for prostate cancer is allocated into an intervention group and a control group. A total of 100 men will be included for a power of 80%. The intervention group will be instructed to use the "Ferticare 2.0" vibrator for at least five minutes a day with an amplitude of 1 mm and frequency of 90 Hz (these settings were found in a pilot study) for a total of 9 months.

Both groups will do the standard pelvic floor training program and both groups will be offered regular phosphodiesterase-5-inhibitor treatment. Before surgery, 3, 6 and 10 months after the patients will have to fill out four different questionnaires regarding sexual and urinary function, including IIEF-EF, EHS, "neglected side effects" and ICIQ-SF. (10 months is due to a wash-out period of 1 month after the intervention).

The collected data will be analysed and the primary goal is to see if there is a significant difference in average spontaneous IIEF-EF score in the two groups 10 months after the surgery.

DETAILED DESCRIPTION:
Hypothesis The study's hypothesis is that vibration therapy, using the stimulation parameters found in the pilot study, will have a beneficial effect on erectile function, orgasm disturbances, penile shortening, and urinary incontinence, both generally and in connection with sexual activity.

Methods The study is conducted as a randomized, controlled non-blinded study. Men undergoing a nerve-sparing operation for prostate cancer are divided into two groups. A total of 100 men will be included in the study. In case a surgery cannot be performed with nerve preservation or if a participant experiences a recurrence of their prostate cancer requiring additional treatment, the participant will be withdrawn from the study.

Randomization and Treatment Overall, we will investigate the effect of vibration stimulation on erectile function, orgasm disturbances, penile shortening, and urinary incontinence, both generally and in connection with sexual activity. In accordance with the hypotheses, this study will offer vibration therapy for a longer duration than before. Both the vibration group and the control group will be offered fixed post-operative treatment with phosphodiesterase-5-inhibitors as per the standard protocol. Participants will be randomized into the two groups through drawing lots for either vibration or no vibration. Randomization will be done using block randomization via a computer-generated list. The "Ferticare 2.0" vibrator (produced by the company Reflexonic LLC, Leesburg VA, USA) will be used in the study, which is a modernized version of the previously used vibrator and is sold as a sexual aid in Denmark. It is safety-approved with European CE marking as a "household appliance" and is sold as a sexual aid in Denmark. Men in the vibration group will be instructed on the stimulation before their prostate surgery. Subsequently, participants will be able to perform the vibration therapy themselves at home. In both groups, participants must undergo a standard pelvic floor training program, and both groups will be offered fixed PDE-5 inhibitor treatment in the form of daily tadalafil, 5 mg, as the standard treatment for erectile difficulties after the operation. In the vibration group, daily stimulation will be directed towards the frenulum for a minimum of 5 minutes, with an amplitude of 1 mm and a frequency of 90 Hz, as found in the pilot study. Participants will start getting used to the vibration 1-4 weeks before the surgery and resume it within 14 days after the operation. The daily stimulation will continue for a period of 9 months, along with the standard treatment. After these 9 months, men in both groups will stop taking tadalafil during a 4-week wash-out period, after which their spontaneous sexual function will be evaluated. This is necessary due to the well-known positive effect of the medication. In comparison to the standard treatment in the department, offering vibration to half of the participants is an addition. Regarding pelvic floor training and medication for erectile difficulties for all study participants, the current standard is to offer these to all men who have undergone nerve-sparing radical prostatectomy. This will proceed as usual, and the only deviation from usual practice is ensuring that the medication offer is consistent for all participants. The mentioned 4-week period without tablet treatment (wash-out) is necessary to assess spontaneous erections. This is a deviation from the normal standard, as such a wash-out is not conducted for patients who do not participate in research, but it will not affect the actual erectile function of the participants in either group.

Data Collection

Standard investigations related to prostate cancer will be conducted according to normal guidelines, with the registration of:

* Pre-operative PSA
* Clinical and pathological tumor stage
* Gleason score
* Prostate size
* Degree of nerve preservation during the surgery
* Any complications during the surgery
* Resection margin status (positive or negative)
* PSA measurements at 3, 6, and 12 months after the operation. This information will be obtained from the patient's medical records by the scientific staff after the study participants have given their consent to participate. After providing consent, the study organizers, sponsor, sponsor's representatives, and any regulatory authorities will have direct access to obtain information from the patient's medical records, including electronic records, for the purpose of reviewing information about the research participant's health, as necessary for conducting the research project and for monitoring, including self-monitoring, quality control, and oversight, as they are obligated to perform.

Since potential participants are screened and informed about the project during their visits to the outpatient clinic (see the section on Recruitment of Study Participants and Informed Consent), there is no need to obtain information from the patient's medical records before consent is given. At this stage, the research team only receives the name, social security number, and contact information for patients who have expressed interest in the project.

Additional examinations are carried out before the surgery and at follow-ups at 3 months, 6 months, and 10 months (equivalent to the end of the wash-out period) after the surgery, with the registration of the following for all participants in both the vibration group and the control group:

Before the surgery and at follow-ups:

* Validated symptom questionnaires for erectile function (IIEF-EF and EHS)
* Specific questionnaire about orgasm disturbances, penile shortening, and urinary incontinence during sexual activity.
* Validated symptom questionnaire for incontinence symptoms (ICIQ-SF)
* 24-hour pad weighing test (only at follow-ups for men who are not fully continent)

Additional registrations at follow-ups:

* Registration of PSA recurrence after the surgery and noting any additional treatment
* Any side effects of vibration and standard treatment

ELIGIBILITY:
Inclusion Criteria:

* Men who are undergoing nerve-sparing radical prostatectomy
* Pre operative erectile function of IIEF-EF > 25
* Sexually active . Continent before surgery defined as a score of 0 on the ICIQ-SF questionnaire

Exclusion Criteria:

* Urinary incontinent before surgery
* Comorbidity that prevents the patient from taking PDE5-inhibitors
* Disease in the penis or in the penile skin (Peyronies, phimosis)
* Problems using the vibrator ie impaired function of the hands

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Erectile function | 10 months
  The erectile function compared to controls measured by IIEF-EF

SECONDARY OUTCOMES:
ICIQ-UI-SF: The International Consultation on Incontinence Questionnaire - Urinary Incontinence - short form | 10 months
  Difference in ICIQ-SF score between the two groups after 3, 6 and 10 months. The score is from 0-21. The higher the score the more incontinent. A score of 0 is no urinary incontinence.
IIEF-EF score (The International Index of Erectile Function - Erectile Function) | 10 months
  Difference in IIEF-EF score between the two groups after 3, 6 and 10 months. The minimum score is 0 and the maximum score is 30. The higher the score the better erectile function.
Diaper weighing test | 10 months
  Difference in 24 hour diaper weighing test between the two groups after 3, 6 and 10 months
IIEF-EF (The International Index of Erectile Function - Erectile Function) over 25 | 10 months
  The percentage of patients who gain a post-operative spontaneous IIEF-EF score of at least 25. The minimum score is 0 and the maximum score is 30. The higher the score the better erectile function.
EHS (Erection Hardness Scale) | 10 months
  The percentage of patients who gain a post-operative spontaneous EHS of at least 3. The scale is from 0-4. 0 is no erection, the higher the score the better erection.
Neglected sexual side effects | 10 months
  The presence of orgasm disturbances, penile shortening and urinary incontinence in relation to sexual activity.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Fode, MD, PhD, Principal Investigator — Department of Urology, Herlev and Gentofte University Hospital
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Available upon request. Subject to approval from the Danish Data Protection Agency.
Supporting Information: Study Protocol, SAP